CLINICAL TRIAL: NCT04639258
Title: Medtronic Evolut™ EXPAND TAVR I Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reevaluation of clinical strategy in this patient population led to a business decision to discontinue the study. Discontinuation is not due to any patient safety, patient welfare, or quality issues.
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D00266108
Record Dates: First submitted 2020-11-05; First posted 2020-11-20 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Medtronic Evolut™ PRO+ System (Experimental): All study subjects will be treated with the Medtronic Evolut™ PRO+ TAVR System.
  Interventions: Device: Medtronic Evolut™ PRO+ System

INTERVENTIONS:
Device: Medtronic Evolut™ PRO+ System — TAVR treatment with Medtronic Evolut™ PRO+ System

SUMMARY:
The purpose of the study is to obtain safety and effectiveness data of the Medtronic Evolut™ PRO+ TAVR System for the treatment of severe, asymptomatic aortic stenosis.

DETAILED DESCRIPTION:
Single-arm, descriptive, multi-center, international

All subjects will be treated with a Medtronic Evolut™ PRO+ TAVR System. Subject follow-ups will be conducted at pre and post-procedure, discharge, 30 days, 6 months, and annually through 5 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Severe aortic stenosis, defined as: Aortic valve area ≤ 1.0 cm^2, or aortic valve area index ≤ 0.6 cm^2/m^2, and mean gradient ≥ 40 mmHg or Vmax ≥ 4.0 m/sec
* Subject denies symptoms attributable to aortic stenosis, including but not limited to:

  * Dyspnea on rest or exertion
  * Angina
  * Syncope in the absence of another identifiable cause
  * Fatigue
  * Left Ventricular Ejection Fraction (LVEF) >50%

Key Exclusion Criteria:

* Age <65 years
* Class I indication for cardiac surgery
* Bicuspid, unicuspid, or quadricuspid aortic valve
* In need of and suitable for coronary revascularization

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sorajja, MD, Principal Investigator — Allina Health System; Josep Rodes-Cabau, MD, Principal Investigator — Fondation IUCPQ
Locations (8):
- United States (4):
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - Northwell Health, Manhasset, New York
  - UPMC Pinnacle Harrisburg Campus, Wormleysburg, Pennsylvania
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- The Alfred Hospital, Melbourne, Australia
- IUCPQ, Québec, Canada
- Rabin Medical Center, Petah Tikva, Israel
- Waikato Hospital, Hamilton, New Zealand

RESULTS

PARTICIPANT FLOW:
Groups:
- TAVR: Up to 75 subjects with moderate, symptomatic AS
Period: Overall Study
Arm/Group | TAVR
Started | 11
Completed | 0
Not Completed | 11
Not completed — Screen failure | 5
Not completed — Physician Decision | 2
Not completed — Early study termination | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: No subject had an attempted TAVR procedure.
  As full baseline data is only required for subjects who are approved for treatment it was not reported for all subjects. No subjects were approved for treatment. Of the 11 enrolled (consented) subjects 8 had baseline data reported.
Groups:
- TAVR: Up to 75 subjects with moderate, symptomatic AS with an attempted TAVR procedure
Arm/Group | TAVR
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 76.9 [68 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 2
  United States | 3
  Australia | 3
NYHA Classification [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Participants
    Class I | 5
    Class II | 0
    Class III | 0
    Class IV | 0
    Unknown/Not Reported | 3
Society of Thoracic Surgeons (STS) Score [Mean (Full Range); unit: Percentage] — Measure Description: Society of Thoracic Surgeons (STS) score of predicted risk of 30-day mortality following surgical aortic valve replacement. The score is measured as a percentage (0-100%) with higher scores representing a higher probability of mortality at 30 days. Population: STS score was reported for 6 participants
  Percentage
    number analyzed (Participants) | 6
    (all) | 2.9 [0.8 to 5.9]
BSA [Mean (Full Range); unit: m^2] — Body surface area reporting in meters squared Population: Body surface area was reported for 6 participants.
  m^2 | 1.7 [1.4 to 1.9]

OUTCOME MEASURES:

1. Primary Outcome: All-cause and Cardiovascular Mortality
Description: Rate of all-cause and cardiovascular mortality
Time Frame: 30 days
Population: No subjects with an attempted TAVR procedure.
  No data is reported as statistical analysis plan specifies that results would be reported for:
  * Attempted Implant (all subjects with an attempted procedure)
  * Implanted (all subjects with an attempted procedure where the study device is implanted)
Arm/Group | TAVR
Number analyzed (Participants) | 0

2. Primary Outcome: All-cause and Cardiovascular Mortality
Description: Rate of all-cause and cardiovascular mortality
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

3. Primary Outcome: All Stroke (Disabling and Non-disabling)
Description: Rate of disabling and non-disabling stroke
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

4. Primary Outcome: All Stroke (Disabling and Non-disabling)
Description: Rate of disabling and non-disabling stroke
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

5. Primary Outcome: Myocardial Infarction (Periprocedural and Spontaneous)
Description: Rate of periprocedural and spontaneous myocardial infarction
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

6. Primary Outcome: Myocardial Infarction (Periprocedural and Spontaneous)
Description: Rate of periprocedural and spontaneous myocardial infarction
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

7. Primary Outcome: Acute Kidney Injury
Description: Rate of acute kidney injury
Time Frame: 30 days
Population: No subjects with an attempted TAVR procedure
  No data is reported as statistical analysis plan specifies that results would be reported for:
  * Attempted Implant (all subjects with an attempted procedure)
  * Implanted (all subjects with an attempted procedure where the study device is implanted)
Arm/Group | TAVR
Number analyzed (Participants) | 0

8. Primary Outcome: Acute Kidney Injury
Description: Rate of acute kidney injury
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

9. Primary Outcome: Major Vascular Complications
Description: Rate of major vascular complications
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

10. Primary Outcome: Major Vascular Complications
Description: Rate of major vascular complications
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

11. Primary Outcome: Life-threatening Bleed
Description: Rate of life-threatening (or disabling) bleed
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

12. Primary Outcome: Life-threatening Bleed
Description: Rate of life-threatening (or disabling) bleed
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

13. Primary Outcome: New Permanent Pacemaker Implantation (PPI)
Description: Rate of new permanent pacemaker implantation (excludes patients with pre-existing pacemakers at baseline)
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

14. Primary Outcome: New Permanent Pacemaker Implantation (PPI)
Description: Rate of new permanent pacemaker implantation (excludes patients with pre-existing pacemakers at baseline)
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

15. Primary Outcome: New Intraventricular Conduction Delays
Description: Rate of new intraventricular conduction delays (excludes patients with intraventricular conduction delays at baseline)
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

16. Primary Outcome: New Intraventricular Conduction Delays
Description: Rate of new intraventricular conduction delays (excludes patients with intraventricular conduction delays at baseline)
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

17. Primary Outcome: New-onset Atrial Fibrillation
Description: Rate of new-onset atrial fibrillation (excludes patients with atrial fibrillation at baseline)
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

18. Primary Outcome: New-onset Atrial Fibrillation
Description: Rate of new-onset atrial fibrillation (excludes patients with atrial fibrillation at baseline)
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

19. Primary Outcome: Valve-related Dysfunction Requiring Repeat Procedure
Description: Rate of valve-related dysfunction requiring repeat procedure
Time Frame: 30 days
Population: Can only be observed following a successful TAVR procedure. Cannot be reported on as there were no subjects with an attempted or successful TAVR procedure.
Arm/Group | TAVR
Number analyzed (Participants) | 0

20. Primary Outcome: Valve-related Dysfunction Requiring Repeat Procedure
Description: Rate of valve-related dysfunction requiring repeat procedure
Time Frame: 6 months
Population: as for outcome 19
Arm/Group | TAVR
Number analyzed (Participants) | 0

21. Primary Outcome: Device Success (VARC-2)
Description: The VARC-2 definition of device success is absence of procedural mortality, correct positioning of a single prosthetic heart valve into the proper anatomical location, intended performance of the prosthetic heart valve, defined as the absence of patient-prosthesis-mismatch and mean aortic valve gradient less than 20 mmHg (or peak velocity <3 m/sec), and absence of moderate or severe prosthetic valve regurgitation
Time Frame: Discharge (12 hours to 7 days post-procedure)
Population: as for outcome 19
Arm/Group | TAVR
Number analyzed (Participants) | 0

22. Primary Outcome: Cardiovascular and Heart Failure Hospitalizations
Description: Rate of cardiovascular and heart failure hospitalizations
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

23. Primary Outcome: Cardiovascular and Heart Failure Hospitalizations
Description: Rate of cardiovascular and heart failure hospitalizations
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

24. Primary Outcome: Heart Failure Events
Description: Rate of heart failure events
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

25. Primary Outcome: Heart Failure Events
Description: Rate of heart failure events
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

26. Primary Outcome: Hemodynamic Performance Metrics (Mean Aortic Gradient) by Doppler Echocardiography
Description: Reporting of prosthetic valve hemodynamic performance by transvalvular mean aortic gradient
Time Frame: Discharge (12 hours to 7 days post-procedure)
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

27. Primary Outcome: Hemodynamic Performance Metrics (Mean Aortic Gradient) by Doppler Echocardiography
Description: Reporting of prosthetic valve hemodynamic performance by transvalvular mean aortic gradient
Time Frame: 30 days
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

28. Primary Outcome: Hemodynamic Performance Metrics (Mean Aortic Gradient) by Doppler Echocardiography
Description: Reporting of prosthetic valve hemodynamic performance by transvalvular mean aortic gradient
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

29. Primary Outcome: Hemodynamic Performance Metrics (Effective Orifice Area) by Doppler Echocardiography
Description: Change in hemodynamic performance metrics by Doppler echocardiography measured by effective orifice area.
Time Frame: Discharge (12 hours to 7 days post-procedure)
Population: Can only be observed following an attempted or successful TAVR procedure. Cannot be reported on as there were no subjects with an attempted or successful TAVR procedure.
Arm/Group | TAVR
Number analyzed (Participants) | 0

30. Primary Outcome: Hemodynamic Performance Metrics (Effective Orifice Area) by Doppler Echocardiography
Description: Change in hemodynamic performance metrics by Doppler echocardiography measured by effective orifice area.
Time Frame: 30 days
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

31. Primary Outcome: Hemodynamic Performance Metrics (Effective Orifice Area) by Doppler Echocardiography
Description: Change in hemodynamic performance metrics by Doppler echocardiography measured by effective orifice area.
Time Frame: 6 months
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

32. Primary Outcome: Hemodynamic Performance Metrics (Degree of Total, Para, and Transvalvular Prosthetic Regurgitation) by Doppler Echocardiography
Description: Reporting of prosthetic valve hemodynamic performance by degree of total, para, and transvalvular regurgitation by Doppler echocardiography
Time Frame: Discharge (12 hours to 7 days post-procedure)
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

33. Primary Outcome: Hemodynamic Performance Metrics (Degree of Total, Para, and Transvalvular Prosthetic Regurgitation) by Doppler Echocardiography
Description: as for outcome 32
Time Frame: 30 days
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

34. Primary Outcome: Hemodynamic Performance Metrics (Degree of Total, Para, and Transvalvular Prosthetic Regurgitation) by Doppler Echocardiography
Description: as for outcome 32
Time Frame: 6 months
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

35. Primary Outcome: Hemodynamic Performance Metrics (Incidence of Moderate and Severe Patient-prosthesis Mismatch) by Doppler Echocardiography
Description: Reporting of prosthetic valve hemodynamic performance by incidence of moderate and severe patient-prosthesis mismatch by Doppler echocardiography
Time Frame: Discharge (12 hours to 7 days post-procedure)
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

36. Primary Outcome: Hemodynamic Performance Metrics (Incidence of Moderate and Severe Patient-prosthesis Mismatch) by Doppler Echocardiography
Description: as for outcome 35
Time Frame: 30 days
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

37. Primary Outcome: Hemodynamic Performance Metrics (Incidence of Moderate and Severe Patient-prosthesis Mismatch) by Doppler Echocardiography
Description: as for outcome 35
Time Frame: 6 months
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

38. Primary Outcome: Change From Baseline in New York Heart Association (NYHA) Functional Classification
Description: Reporting of NYHA classification change from baseline to 30 days and 6 months
  NYHA Classification criteria:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
Time Frame: 30 days and 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

39. Primary Outcome: Change From Baseline in Six-minute Walk Test (6MWT)
Description: Reporting change from baseline in distance walked during 6MWT
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

40. Primary Outcome: Change From Baseline in Health-related Quality of Life (QoL) as Assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: KCCQ quantifies physical function, symptoms, social function, self-efficiency, knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: 30 days and 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

41. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Description: Reporting of change in left ventricular ejection fraction (LVEF) from baseline by echocardiography
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

42. Primary Outcome: Change From Baseline in Global Longitudinal Strain (GLS)
Description: Reporting of change in GLS from baseline by echocardiography
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

43. Primary Outcome: Change From Baseline in Left Ventricular Filling Pressure (E:e')
Description: Reporting of change in left ventricular filling pressure (E:e') from baseline by echocardiography
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

44. Primary Outcome: Change From Baseline in Stroke Volume Index (SVI)
Description: Reporting of change in stroke volume index (SVI) from baseline by echocardiography
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

45. Primary Outcome: Change From Baseline in NT-pro B-type Natriuretic Peptide (NT-proBNP)
Description: Reporting of change in NT-pro B-type natriuretic peptide (NT-proBNP) from baseline
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

46. Other Pre Specified Outcome: All-cause and Cardiovascular Mortality
Description: Rate of all-cause and cardiovascular mortality
Time Frame: Annually through 5 years
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

47. Other Pre Specified Outcome: All Stroke (Disabling and Non-disabling)
Description: Rate of disabling and non-disabling strokes
Time Frame: Annually through 5 years
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

48. Other Pre Specified Outcome: Cardiovascular and Heart Failure Hospitalizations
Description: Rate of cardiovascular and heart failure hospitalizations
Time Frame: Annually through 5 years
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

49. Other Pre Specified Outcome: Heart Failure Events
Description: Rate of heart failure events
Time Frame: Annually through 5 years
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

50. Other Pre Specified Outcome: New York Heart Association (NYHA) Functional Classification
Description: Reporting NYHA functional classification by timepoint following attempted procedure
Time Frame: 30 days, 6 months, and annually through 5 years
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

51. Other Pre Specified Outcome: Change From Baseline in New York Heart Association (NYHA) Functional Classification
Description: as for outcome 38
Time Frame: Annually through 5 years
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

52. Other Pre Specified Outcome: Health-related Quality of Life (QoL) as Assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: as for outcome 40
Time Frame: Annually through 5 years
Population: as for outcome 1
Arm/Group | TAVR
Number analyzed (Participants) | 0

53. Other Pre Specified Outcome: Hemodynamic Performance Metrics (Mean Aortic Gradient) by Doppler Echocardiography
Description: Reporting of prosthetic valve hemodynamic performance by transvalvular mean aortic gradient
Time Frame: Annually through 5 years
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

54. Other Pre Specified Outcome: Hemodynamic Performance Metrics (Effective Orifice Area) by Doppler Echocardiography
Description: Reporting of prosthetic valve hemodynamic performance by effective orifice area (EOA)
Time Frame: Annually through 5 years
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

55. Other Pre Specified Outcome: Hemodynamic Performance Metrics (Degree of Total, Para, and Transvalvular Prosthetic Regurgitation) by Doppler Echocardiography
Description: Reporting of prosthetic valve hemodynamic performance by degree of total, para, and transvalvular prosthetic regurgitation by Doppler echocardiography
Time Frame: Annually through 5 years
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

56. Other Pre Specified Outcome: Hemodynamic Performance Metrics (Incidence of Moderate and Severe Patient-prosthesis Mismatch) by Doppler Echocardiography
Description: as for outcome 35
Time Frame: Annually through 5 years
Population: as for outcome 29
Arm/Group | TAVR
Number analyzed (Participants) | 0

57. Other Pre Specified Outcome: Prosthetic Valve Thrombosis
Description: Rate of prosthetic valve thrombosis
Time Frame: 30 days, 6 months, and annually through 5 years
Population: as for outcome 19
Arm/Group | TAVR
Number analyzed (Participants) | 0

58. Other Pre Specified Outcome: Prosthetic Valve Endocarditis
Description: Rate of prosthetic valve endocarditis
Time Frame: 30 days, 6 months, and annually through 5 years
Population: as for outcome 19
Arm/Group | TAVR
Number analyzed (Participants) | 0

59. Other Pre Specified Outcome: Bioprosthetic Valve Dysfunction (BVD)
Description: Rate of bioprosthetic valve dysfunction (BVD)
Time Frame: 30 days, 6 months, and annually through 5 years
Population: as for outcome 19
Arm/Group | TAVR
Number analyzed (Participants) | 0

60. Other Pre Specified Outcome: Bioprosthetic Valve Failure (BVF)
Description: Rate of bioprosthetic valve failure (BVF)
Time Frame: 30 days, 6 months, and annually through 5 years
Population: as for outcome 19
Arm/Group | TAVR
Number analyzed (Participants) | 0

61. Other Pre Specified Outcome: Valve-related Dysfunction Requiring Repeat Procedure
Description: Rate of valve-related dysfunction requiring repeat procedure
Time Frame: Annually through 5 years
Population: as for outcome 19
Arm/Group | TAVR
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from study enrollment (consent) through study exit, up to 151 days. First subject was enrolled on 28 May 2021 and last subject was exited on 28 Feb 2022. No study subjects were treated. If subjects had been treated all AEs would have been reported through 6 months post-procedure. After 6 months post-procedures only serious adverse events, device-related events, and device deficiencies would have been reported.
Description: The definitions used for AEs and SAEs is too long for the field. The definitions differed in that the CIP used the definitions found in ISO14100:2020.
  Investigators are required to evaluate and document in the subject's medical records all adverse events and device deficiencies observed in study subjects from the time they are enrolled until they are exited from the study. All AEs should be followed through their resolution.
Arm/Group | TAVR
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR (N=11)
Coronary stenosis (Cardiac disorders) | 1 (1)
Left radial artery pseudoaneurysm following study specific angiogram (Injury, poisoning and procedural complications) | 1 (1)
Haematome, left radial (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR (N=11)
Scalp laceration (Injury, poisoning and procedural complications) | 1 (1)
Parasthesia, left thumb and index finger (Nervous system disorders) | 1 (1)
Bilateral ovarian cysts (Reproductive system and breast disorders) | 1 (1)
Saccular infrarenal abdominal aortic aneurysm (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of the study prior to any attempted TAVR procedures led to no evaluable subjects for data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 60 days of receipt Medtronic (MDT) will verify presence of Confidential Information (CI) & won't censor or interfere with presentation/conclusions except to protect CI (other than Study Data) & its rights in patentable or copyrightable materials, & check technical accuracy of MDT data. If told by MDT that Publication contains CI or technical errors of MDT data, PI will make requested changes before publishing/presenting. PI will delay publication up to 90 more days, if requested.

DOCUMENTS (2):
  • Study Protocol (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT04639258/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT04639258/SAP_002.pdf